CLINICAL TRIAL: NCT06184438
Title: Randomized Control Trial of Micronized Purified Flavonoid Fraction for Post Operative Treatment in Anal Fistula Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Principal Investigator, Tungcheng Chang, MD, PhD, Chief of Colorectal Surgery, Taipei Medical University Shuang Ho Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N202309013
Record Dates: First submitted 2023-12-14; First posted 2023-12-28 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Anal Fistula
Keywords: flavnoids; fistulotomy; fistulectomy
MeSH Terms: conditions — Rectal Fistula | interventions — Diosmin; Hesperidin; Control Groups

STUDY DESIGN:
Intervention Model Description: We designed a randomized controlled trial including 150 eligible patients who underwent fistulotomy or fistulectomy. To evaluate the benefit of using MPFF after fistula surgery, patients were classified into 2 groups:
  1. Received MPFF(Daflon 1000mg BID) after surgery.
  2. Received placebo after surgery.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Daflon group (Experimental): Received Micronized purified flavonoid fraction(Daflon 1000mg) BID after surgery from day 0 to day 7.
  Interventions: Drug: Micronized purified flavonoid fraction(Daflon 1000mg)
- Placebo group (Placebo Comparator): Received placebo after surgery from day 0 to day 7.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Micronized purified flavonoid fraction(Daflon 1000mg) — Received Micronized purified flavonoid fraction(Daflon 1000mg) BID after surgery from day to day 7
  Other Names: diosmin; hesperidin
  Arms: Daflon group
Drug: Placebo — Received placebo after surgery.
  Other Names: Control group
  Arms: Placebo group

SUMMARY:
The aim of this study is to evaluate the effect of micronized purified flavonoid fraction on postoperative symptoms after surgery of anorectal fistulas.

DETAILED DESCRIPTION:
The current theory of cryptoglandular suggest that perianal fistula occurs when the anal crypt glands become occluded and infected, over 90% of perianal fistulas are cryptoglandular in origin and arise from perianal abscesses. Also inflammatory process might play an important role in the formation of cryptoglandular perianal fistula. This condition is mainly managed with surgery, currently remain majorly on two conventional surgical interventions--fistulotomy and fistulectomy.

MPFF is a drug to treat venous vessel disease such as varicose and hemorrhoid, which was found with effects of lowering lymphatic permeability, improving venous return and vessel endothelial inflammation. More research has also shown the effects of MPFF on post hemorrhoidectomy symptom control, such as bleeding, pain, and infection. Since other anorectal surgery has similar complications. Therefor we conducted this randomized control trial to evaluate the benefits of MPFF after anal fistula surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo fistulectomy or fistulotomy are included.

Exclusion Criteria:

* Emergency operation
* Participants who had Trans-sphincteric anal fistula, Extra-sphincteric anal fistula
* Participants accompanied by severe liver cirrhosis
* Participants accompanied by coagulation disorders
* Participants taking anticoagulant
* Participants taking corticosteroids as long-term medication.
* Participants who had colorectal cancer
* Participants taking analgesic drugs (morphine or others) as long-term medication
* Participants bed-ridden
* Participants who had history of human immunodeficiency virus (HIV) infection
* Pregnant woman

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2023-12-13 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Post-operative pain | 0-7 days
  Record the maximum pain score(visual analog scale, 0-10) from post-operative day 0 to day 7.
Frequency of dressing replacement | 0-7 days
  Record the frequency of dressing replacement from post-operative day 0 to day 7.

SECONDARY OUTCOMES:
Analgesic agent use | 0-7days
  Daily consumption of oral analgesics from post-operative day 0 to day 7
Incidence of surgical site infection | 0-30 days
  Surgical site infection was defined as hospital admission for infection management or need for surgical intervention to manage the wound.
Incidence of urinary retention | 0-7days
  Urinary retention was defined as patients requiring Foley catheterization during the hospital stay.
Daily activity | 0-7 days
  The number of days the patient takes to go back to work.
Bowel movement | 0-7 days
  Duration until first bowel movement after surgery.
Patient satisfaction | Post Operative day 7
  Questionnaire will be collected after the surgery.
Length of hospital stay | 0-7 days
  Length of hospital stay after the surgery.
Wound healing questionnaire | 0-60 days
  Evaluate wound healing at 30 days after operation.

CONTACTS AND LOCATIONS:
Overall Officials: Tungcheng Chang, MD, PHD, Study Director — Taipei Medical University Shuang Ho Hospital
Locations (1):
- Taipei Medical University Shuang-Ho Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
The datasets used in this study can be obtained from the investigator upon reasonable request.
Supporting Information: Study Protocol
Time Frame: data is available as the study is complete and for 12 month period
Access Criteria: will be shared upon request